CLINICAL TRIAL: NCT07365397
Title: Comparative Study on Imaging Characteristics of Different ⁶⁸Ga-Labeled PSMA Probes in Patients With Prostate Cancer
Brief Title: Imaging Characteristics of Different ⁶⁸Ga-PSMA Probes in Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GenSciP153-001
Record Dates: First submitted 2026-01-14; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 68Ga-GS24-B2-250-T (Experimental): detect prostate cancer lesions via 68Ga-GS24-B2-250-T PET/CT imaging
  Interventions: Diagnostic Test: 68Ga-GS24-B2-250-T; Diagnostic Test: 68Ga-PSMA-11
- 68Ga-GS24-B2-237-T (Experimental): detect prostate cancer lesions via 68Ga-GS24-B2-237-T PET/CT imaging
  Interventions: Diagnostic Test: 68Ga-GS24-B2-237-T; Diagnostic Test: 68Ga-PSMA-11
- 68Ga-GS24-B2-268-T (Experimental): detect prostate cancer lesions via 68Ga-GS24-B2-268-T PET/CT imaging
  Interventions: Diagnostic Test: 68Ga-GS24-B2-268-T; Diagnostic Test: 68Ga-PSMA-11

INTERVENTIONS:
Diagnostic Test: 68Ga-GS24-B2-268-T — detect prostate cancer lesions via 68Ga-GS24-B2-268-T PET/CT imaging
  Arms: 68Ga-GS24-B2-268-T
Diagnostic Test: 68Ga-GS24-B2-250-T — detect prostate cancer lesions via 68Ga-GS24-B2-250-T PET/CT imaging
  Arms: 68Ga-GS24-B2-250-T
Diagnostic Test: 68Ga-GS24-B2-237-T — detect prostate cancer lesions via 68Ga-GS24-B2-237-T PET/CT imaging
  Arms: 68Ga-GS24-B2-237-T
Diagnostic Test: 68Ga-PSMA-11 — detect prostate cancer lesions via 68Ga-PSMA-11 PET/CT imaging

SUMMARY:
This study aims to evaluate the imaging characteristics of [⁶⁸Ga]Ga-GS24-B2-250-T Injection (abbreviated as ⁶⁸Ga-GS24-B2-250-T), [⁶⁸Ga]Ga-GS24-B2-268-T Injection (abbreviated as ⁶⁸Ga-GS24-B2-268-T), [⁶⁸Ga]Ga-GS24-B2-237-T Injection (abbreviated as ⁶⁸Ga-GS24-B2-237-T), and [⁶⁸Ga]Ga-PSMA-11 Injection (abbreviated as ⁶⁸Ga-PSMA-11) as PET/CT imaging agents in patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has fully understood the trial content, process, and potential risks, and has voluntarily signed the informed consent form;
2. Male subjects aged ≥ 18 years;
3. Clinically or radiologically assessed as metastatic hormone-sensitive prostate cancer (mHSPC) or metastatic castration-resistant prostate cancer (mCRPC);
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
5. Presence of positive lesions on ⁶⁸Ga-PSMA-11 PET/CT scan;
6. Blood routine, renal function, and liver function tests meeting the following criteria:

   1. Platelet count > 90 × 10⁹/L;
   2. Urea/urea nitrogen and serum creatinine < 1.5 × upper limit of normal (ULN);
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 × ULN;
7. Expected survival time ≥ 6 months;
8. From the date of signing the informed consent form until 3 months after administration, the subject and his partner must use effective contraceptive measures, and the subject must avoid sperm donation.

Exclusion Criteria:

1. Having participated in another interventional clinical trial prior to signing the informed consent form and being within 5 half-lives of the investigational product of that trial; or currently participating in another interventional clinical trial; or having participated in a clinical trial involving radiopharmaceuticals prior to signing the informed consent form with an interval of less than 3 months between the last dose and the informed consent signing date.
2. Having received any intravenous iodine-containing contrast agent within 24 hours prior to administration, or any high-density oral contrast agent (e.g., barium sulfate) within 5 days prior to administration. Oral water-soluble contrast agents (e.g., compound meglumine diatrizoate oral solution) are acceptable.
3. Having received high-energy γ-ray-emitting agents (>300 KeV, e.g., radiopharmaceuticals labeled with radionuclides such as [¹³¹I]I, [¹⁸F]F, [⁶⁸Ga]Ga, [⁶⁴Cu]Cu, etc.) within a period equivalent to either 5 half-lives of the agent or 2 days, whichever is longer, prior to administration.
4. Planning to adjust anti-tumor medication during the study period.
5. Being unable to complete the required PET/CT imaging procedures.
6. Having any medical condition or other circumstances that, in the investigator's judgment, may affect the safety or compliance of the subject.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-07-26 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Value for major organs (salivary glands, kidneys, bone marrow, etc.) and tumor lesions (primary and metastatic lesions) | 5 days
  The Standardized Uptake Value (SUVmax and SUVmin) of major organs (salivary glands, kidneys, bone marrow, etc) and tumor lesions (primary and metastatic lesions) is measured by using Positron Emission Tomography/Computed Tomography (PET/CT) imaging technology for both 68Ga-PSMA-11 and other tested tracers.

IPD SHARING:
Plan to Share IPD: No